CLINICAL TRIAL: NCT00325663
Title: Specific and Non-Specific Effects of Acupuncture: A Double-Blinded, Randomized, Controlled Trial in Patients With Osteoarthritis of the Knee
Brief Title: Acupuncture in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: The German Society for Traditional Chinese Medicine (DGTCM) (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AKOK1
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2004-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: acupuncture; double-blind; sham control; osteoarthritis; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The aim of this study was to evalute three different acupuncture techniques, including one sham control, in its effect on osteoarthitis of the knee

DETAILED DESCRIPTION:
Background: Acupuncture is one of the most frequently used complementary therapeutic approaches in the treatment of osteoarthritis of the knee. Due to methodological shortcomings of previous randomized controlled studies, controversy persists whether the observed effects are specific to acupuncture or non-specific consequences of needling.

Objective: To compare classical Chinese acupuncture, semi-standardized modern acupuncture and non-specific needling by means of a double-blinded repeated measures cross-over design.

Intervention: Within three weeks all patients receive three treatment modalities in a random order in a double-blind study design.

Main outcome measures: Improvement in knee flexibility according to the neutral-zero method, defining a success as improvement by 10 degrees or more.

Secondary parameter: improvement in pain according to the reduced WOMAC score by 50 percent or more.

ELIGIBILITY:
Inclusion Criteria:

* Patients above age 35
* knee osteoarthritis grade II or III according to the Kellgren classification.

Exclusion Criteria:

* orthopedic deformations of the knee,
* malignant disease
* auto-immune disorders
* surgery including arthroscopy during the past 12 months
* pain medication with steroids
* physical therapy or acupuncture within the last for weeks
* no or a pain medication in continuous dosage

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2004-04; Study Completion 2005-04

PRIMARY OUTCOMES:
Main outcome measures: Improvement in knee flexibility according to the neutral-zero method, defining a success as improvement by 10 degrees or more.

SECONDARY OUTCOMES:
Secondary parameter: improvement in pain according to the reduced WOMAC score by 50 percent or more.

CONTACTS AND LOCATIONS:
Overall Officials: Max Karner, MD, Principal Investigator — University Heidelberg; Johannes Greten, MD, Study Director — German Society of Traditional Chinese Medicine; Oliver Gerlach, MD, Study Chair — Shen-Centre for Traditional Chinese Medicine, Erlangen, Germany; Frank Brazkiewicz, MD, Study Chair — Centre for Chinese Medicine, Bremen, Germany